CLINICAL TRIAL: NCT02734940
Title: Multimodal Analgesia in Cardiac Surgery (Pilot Study)
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Unable to find participants who met inclusion/exclusion criteria
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HM20004692
Record Dates: First submitted 2016-03-09; First posted 2016-04-12 (Estimated); Results first posted 2018-02-19 (Actual); Last update posted 2018-08-07 (Actual); Status verified 2018-07

CONDITIONS: Heart Diseases
MeSH Terms: conditions — Heart Diseases | interventions — Lidocaine; Ketamine; Dexmedetomidine; Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Unrestricted Fentanyl (Active Comparator): Will receive injection of sterile saline (2cc) in lower back area (to minimize participant bias) and unrestricted amount of intraoperative opioids (fentanyl) at the discretion of the Anesthesiologist.
  Both groups will receive General Anesthesia with volatile agents and single dose of iv Tylenol intraoperatively. Both groups of patients will be transported to Intensive Care Unit (ICU) on Dexmedetomidine (dose range 0.25 - 0.7 mcg/kg/hr). Dose titration is based on sedation level and hemodynamic goals set by Cardiac Anesthesiologist.
  Interventions: Drug: Unrestricted Fentanyl
- Lidocaine, Dexmedetomidine and Ketamine (Experimental): Will receive pre-operative spinal duramorph (4mcg/kg up to max dose of 300mcg), intra-operative intravenous (iv) infusion of Ketamine (0.4 mg/kg/hr), Lidocaine (20 mcg/kg/min) and Dexmedetomidine (0.25 mcg/kg/hr) started after induction of General Anesthesia and maintained through the Cardiopulmonary Bypass (CPB) towards the end of surgery. At this point all infusions will be turned off except Dexmedetomidine. The total intraoperative fentanyl dose will be limited to <250mcg (or 3mcg/kg) and total midazolam to ≤ 2mg in the study group.
  Interventions: Drug: Lidocaine; Drug: Ketamine; Drug: Precedex; Drug: Duramorph

INTERVENTIONS:
Drug: Lidocaine — This model would use a combination of intravenous (Dexmedetomidine, Ketamine, Lidocaine) and Spinal (Morphine) drugs.
  Other Names: IV Lidocaine
  Arms: Lidocaine, Dexmedetomidine and Ketamine
Drug: Unrestricted Fentanyl — No changes to current practices, using unlimited narcotic medications intraoperatively.
  Other Names: Unlimited intraoperative opiates
  Arms: Unrestricted Fentanyl
Drug: Ketamine — This model would use a combination of intravenous (Dexmedetomidine, Ketamine, Lidocaine) and Spinal (Morphine) drugs.
  Arms: Lidocaine, Dexmedetomidine and Ketamine
Drug: Precedex — This model would use a combination of intravenous (Dexmedetomidine, Ketamine, Lidocaine) and Spinal (Morphine) drugs.
  Other Names: IV Precedex
  Arms: Lidocaine, Dexmedetomidine and Ketamine
Drug: Duramorph — This model would use a combination of intravenous (Dexmedetomidine, Ketamine, Lidocaine) and Spinal (Morphine) drugs.
  Other Names: Spinal Duramorph
  Arms: Lidocaine, Dexmedetomidine and Ketamine

SUMMARY:
The investigators objective is to assess the effectiveness of an opioid sparing multimodal approach for enhancing the recovery in Cardiac Surgical patients. This model would use a combination of intravenous (Dexmedetomidine, Ketamine, Lidocaine) and Spinal (Morphine) drugs.

DETAILED DESCRIPTION:
Cardiac surgery is associated with significant acute pain and a proportion of these patients will develop chronic pain.

Opioids are the main stay of analgesia in cardiac surgery because of the safer hemodynamic profile and sedation. However high dose narcotic use is associated with a variety of unwanted side effects prolonging postoperative recovery. There is growing evidence for the effectiveness of multimodal approach utilizing opiate sparing techniques for enhancing patient recovery following surgery. Early extubation has been associated with improved patient outcome and cost effectiveness in cardiac surgery. The investigators objective is to assess the effectiveness of an opioid sparing multimodal approach for enhancing the recovery in Cardiac Surgical patients. This model would use a combination of intravenous (Dexmedetomidine, Ketamine, Lidocaine) and Spinal (Morphine) drugs. All of the above anesthetic drugs have opioid sparing effect in surgical Patients.

Dexmedetomidine use has been associated with decreased cardiac arrhythmias and improved neurological outcome in cardiac surgical patients. Ketamine has been linked with attenuation of postoperative cognitive dysfunction after cardiac surgery. Both intravenous lidocaine and spinal morphine have been shown to reduce opioid consumption in the perioperative period.

ELIGIBILITY:
Inclusion Criteria:

* Elective CABGs and/or Valve replacements, ≥ 18 years old

Exclusion Criteria:

* Re-do cardiac surgery, Acute endocarditis, Circulatory arrest, Emergent cases, Shock, Left Ventricular Assist Device, Transplantation, Transcatheter Aortic Valve Replacement, contraindications for Spinal including coagulopathy and Clopidogrel <7days, psychosis, known allergy to any of the study drugs, Preoperative liver dysfunction (AST/ALT > 2 times normal) and Renal dysfunction (Cr > 2 mg/dL), inability to administer spinal anesthetic, preoperative opioid use, patients who are unable to give their own consent, expected prolonged intubation postoperatively (>12 hrs), prisoners, pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2016-07-11 (Actual); Primary Completion 2017-02-01 (Actual); Study Completion 2017-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Praveen Prasanna, MD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was terminated because of lack of enrollment. No data was ever collected.
Groups:
- Unrestricted Fentanyl: Will receive injection of sterile saline (2cc) in lower back area (to minimize participant bias) and unrestricted amount of intraoperative opioids (fentanyl) at the discretion of the Anesthesiologist.
  Both groups will receive General Anesthesia with volatile agents and single dose of iv Tylenol intraoperatively. Both groups of patients will be transported to Intensive Care Unit (ICU) on Dexmedetomidine (dose range 0.25 - 0.7 mcg/kg/hr). Dose titration is based on sedation level and hemodynamic goals set by Cardiac Anesthesiologist.
  Unrestricted Fentanyl: No changes to current practices, using unlimited narcotic medications intraoperatively.
Period: Overall Study
Arm/Group | Unrestricted Fentanyl | Lidocaine, Dexmedetomidine and Ketamine
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The study was terminated because of lack of enrollment. No data was collected.
Groups:
- Total: Total of all reporting groups
Arm/Group | Unrestricted Fentanyl | Lidocaine, Dexmedetomidine and Ketamine | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical
Sex: Female, Male
Race (NIH/OMB)

OUTCOME MEASURES:

1. Primary Outcome: Pain Scores - Numerical Rating Scale, 0-10
Description: Pain scores recorded 24 hours post extubation by acute pain services nurses (who will be blinded)
Time Frame: 24 hours
Population: The study was terminated because of lack of enrollment. No data was collected.
Arm/Group | Unrestricted Fentanyl | Lidocaine, Dexmedetomidine and Ketamine
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Postoperative Opioid Consumption
Description: Opioid consumption measured in oral morphine equivalents
Time Frame: 24 hours, 48 hours, 72 hours
Population: The study was terminated because of lack of enrollment. No data was collected.
Arm/Group | Unrestricted Fentanyl | Lidocaine, Dexmedetomidine and Ketamine
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Patient Satisfaction
Description: Patient Satisfaction with pain management in first 24 hours post extubation - as measured by acute pain service nurses (who will be blinded)
Time Frame: 24 hours, 48 hours, 72 hours, 7 days, 30 days
Population: The study was terminated because of lack of enrollment. No data was collected.
Arm/Group | Unrestricted Fentanyl | Lidocaine, Dexmedetomidine and Ketamine
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Extubation
Description: Time from arrival to ICU to extubation
Time Frame: Hours from arrival to ICU to endotracheal extubation (maximum of 12 hours)
Population: The study was terminated because of lack of enrollment. No data was collected.
Arm/Group | Unrestricted Fentanyl | Lidocaine, Dexmedetomidine and Ketamine
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: ICU Length of Stay
Time Frame: Days from arrival to ICU to transfer to step down or floor level of care (maximum of 30 days)
Population: The study was terminated because of lack of enrollment. No data was collected.
Arm/Group | Unrestricted Fentanyl | Lidocaine, Dexmedetomidine and Ketamine
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Delirium Scores
Description: CAM-ICU scores at above time points
Time Frame: 24, 48 and 72 hours
Population: The study was terminated because of lack of enrollment. No data was collected.
Arm/Group | Unrestricted Fentanyl | Lidocaine, Dexmedetomidine and Ketamine
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Ionotropic Requirement
Description: Total amount ionotropes required
Time Frame: Total amount ionotropes required intraoperatively (mcg); total amount ionotropes required from time of admission to ICU postoperatively to discharge from hospital (maximum 30 days)
Population: The study was terminated because of lack of enrollment. No data was collected.
Arm/Group | Unrestricted Fentanyl | Lidocaine, Dexmedetomidine and Ketamine
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Bowel Function
Description: Bowel Function
Time Frame: Will determine each day postoperatively if patient has had a bowel movement, measured in days (maximum 30 days)
Population: The study was terminated because of lack of enrollment. No data was collected.
Arm/Group | Unrestricted Fentanyl | Lidocaine, Dexmedetomidine and Ketamine
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Ionotropic Requirement
Description: Total duration of ionotropic requirement (hours)
Time Frame: Total duration ionotropes intraoperatively (hours); total amount ionotropes required from time of admission to ICU postoperatively to discharge from hospital (hours), (maximum 30 days)
Population: The study was terminated because of lack of enrollment. No data was collected.
Arm/Group | Unrestricted Fentanyl | Lidocaine, Dexmedetomidine and Ketamine
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: No data was collected because no participants started the study.
Description: The study was terminated because of lack of enrollment.
Arm/Group | Unrestricted Fentanyl | Lidocaine, Dexmedetomidine and Ketamine
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-13): https://cdn.clinicaltrials.gov/large-docs/40/NCT02734940/Prot_SAP_000.pdf